CLINICAL TRIAL: NCT01592864
Title: A Clinical Study Investigating the Efficacy of a Dentifrice in Providing Long Term Relief From Dentinal Hypersensitivity
Brief Title: The Efficacy of a Dentifrice in Providing Relief From the Pain of Dentinal Hypersensitivity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RH01325
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Results first posted 2014-03-10 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2013-12

CONDITIONS: Dentine Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Tin Fluorides; fluorophosphate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Dentifrice containing stannous fluoride
  Interventions: Drug: Stannous Fluoride
- Arm 2 (Active Comparator): Marketed dentifrice containing Sodium Monofluorophosphate
  Interventions: Drug: Sodium Monofluorophosphate

INTERVENTIONS:
Drug: Stannous Fluoride — dentifice
  Arms: Arm 1
Drug: Sodium Monofluorophosphate — dentifrice
  Arms: Arm 2

SUMMARY:
A study to compare the efficacy of a test dentifrice against a control dentifrice in reducing dentinal hypersensitivity over an eight week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who suffer from tooth sensitivity

Inclusion Criteria:

- none

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- BioSci Research America, Inc., Las Vegas, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: Of 122 participants screened, 2 participants did not meet the study criteria, and 2 withdrew consent before randomization. 118 participants were randomized to study treatments.
Groups:
- Stannous Fluoride (SnF) Dentifrice: Participants brushed whole mouth with 1-inch strip of the test dentifrice 0.454% SnF for one timed minute, ensuring that they brushed all sensitive areas of their teeth. This was followed by rinsing with 5 milliliter (mL) of water.
- Sodium Monofluorophosphate (NaMFP) Dentifrice: Participants brushed whole mouth with 1-inch strip of the control dentifrice (0.76% NaMFP) for one timed minute, ensuring that they brushed all sensitive areas of their teeth. This was followed by rinsing with 5 mL of water.
Period: Overall Study
Arm/Group | Stannous Fluoride (SnF) Dentifrice | Sodium Monofluorophosphate (NaMFP) Dentifrice
Started | 60 | 58
Completed | 60 | 57
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- SnF Dentifrice: Participants brushed whole mouth with 1-inch strip of the test dentifrice containing 0.454% SnF for one timed minute, ensuring that they brushed all sensitive areas of their teeth. This was followed by rinsing with 5 mL of water.
- NaMFP Dentifrice: Participants brushed whole mouth with 1-inch strip of the control dentifrice containing 0.76% NaMFP for one timed minute, ensuring that they brushed all sensitive areas of their teeth. This was followed by rinsing with 5 mL of water.
- Total: Total of all reporting groups
Arm/Group | SnF Dentifrice | NaMFP Dentifrice | Total
Number analyzed (Participants) | 60 | 58 | 118
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.9 (10.9) | 35.5 (10.6) | 36.2 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 37 | 83
  Male | 14 | 21 | 35

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Evaporative Air Sensitivity Pain Response on a Schiff Sensitivity Scale at Week 8
Description: Response to a constant jet of air applied to hypersensitive teeth is evaluated using a Schiff Sensitivity pain response scale. According to this analog scale, pain response for each individual stimulated tooth ranged from 0 to 3; 0 - participant does not respond to air stimulation, 1 - participant responds to air stimulus but does not request discontinuation of stimulus, 2 - participant responds to air stimulus and request discontinuation of stimulus, 3 - participant responds to air stimulus, considers stimulus to be painful and request discontinuation of stimulus.
Time Frame: Baseline to 8 weeks post administration of study treatment
Population: Intent to Treat (ITT) Population: All randomized participants, who were administered with at least one study treatment during the study and provided at least one post-baseline assessment of efficacy. Missing values were not imputed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SnF Dentifrice | NaMFP Dentifrice
Number analyzed (Participants) | 60 | 58
Score on a scale | -0.9 (0.68) | -0.5 (0.44)
Statistical Analysis 1: Comparison: SnF Dentifrice vs NaMFP Dentifrice; Null hypothesis considered change from baseline to be same for both treatments; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment made for multiple comparisons, as primary comparison was pre-specified; ANCOVA with treatment as fixed factor and baseline Schiff Score as covariate; Adjusted Mean Difference = -0.4, 95% CI 2-sided [-0.6 to -0.2] — Difference is 0.454% SnF minus 0.76% NaMFP such that a negative difference favours first named treatment

2. Secondary Outcome: Mean Change From Baseline in Evaporative Air Sensitivity Pain Response on a Schiff Sensitivity Scale at Week 4
Description: Response to a constant jet of air applied to hypersensitive teeth was evaluated using a Schiff Sensitivity pain response scale. According to this analog scale, pain response for each individual stimulated tooth ranged from 0 to 3; 0 - participant does not respond to air stimulation, 1 - participant responds to air stimulus but does not request discontinuation of stimulus, 2 - participant responds to air stimulus and request discontinuation of stimulus, 3 - participant responds to air stimulus, considers stimulus to be painful and request discontinuation of stimulus.
Time Frame: Baseline to 4 weeks post administration of study treatment
Population: ITT Population: All randomized participants, who were administered with at least one study treatment during the study and provided at least one post-baseline assessment of efficacy. Missing values were not imputed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SnF Dentifrice | NaMFP Dentifrice
Number analyzed (Participants) | 60 | 58
Score on a scale | -0.7 (0.58) | -0.2 (0.43)
Statistical Analysis 1: Comparison: SnF Dentifrice vs NaMFP Dentifrice; Null hypothesis considered change from baseline to be same for both treatments; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment made for multiple comparisons, as primary comparison was pre-specified; ANCOVA with treatment as fixed factor and baseline Schiff Score as covariate; Adjusted Mean Difference = -0.4, 95% CI 2-sided [-0.6 to -0.3] — Difference is 0.454% SnF minus 0.76% NaMFP such that a negative difference favours first named treatment

3. Secondary Outcome: Adjusted Mean Change From Baseline in Tactile Sensitivity Pain Response at Week 8
Description: Response to increasing force on hypersensitive teeth was evaluated using a Yeaple Probe pain response scale. The constant pressure probe allowed the examiner to vary the force applied to the dentin surface from 10 grams (g) to an upper threshold of 80 g, in increments of 10g since the values below represents adjusted mean change in baseline, the value can fall below scale range. The greater the pressure the subject was able to tolerate, the less. Change from baseline in tactile response to Week 8 was calculated.
  sensitive the tooth. According to this tactile sensitivity assessment, an increasing force was applied to hypersensitive tooth until a yes response is recorded or the maximum force has been reached.
Time Frame: Baseline to 8 weeks post administration of study treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | SnF Dentifrice | NaMFP Dentifrice
Number analyzed (Participants) | 60 | 58
grams | 21.3 (21.80) | 4.2 (6.18)
Statistical Analysis 1: Comparison: SnF Dentifrice vs NaMFP Dentifrice; Null hypothesis considered change from baseline to be same for both treatments; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment made for multiple comparisons, as primary comparison was pre-specified; ANCOVA with treatment as fixed factor and baseline Schiff Score as covariate; Adjusted Mean Difference = 16.9, 95% CI 2-sided [11.1 to 22.8] — Difference is 0.454% SnF minus 0.76% NaMFP such that a positive difference favours first named treatment

4. Secondary Outcome: Adjusted Mean Change From Baseline in Tactile Sensitivity Pain Response at Week 4
Description: Response to increasing force on hypersensitive teeth was evaluated using a Yeaple Probe pain response scale. The constant pressure probe allowed the examiner to vary the force applied to the dentin surface from 10g to an upper threshold of 80g, in increments of 10g. The greater the pressure the subject was able to tolerate, the less sensitive the tooth. According to this tactile sensitivity assessment, an increasing force was applied to hypersensitive tooth until a yes response is recorded or the maximum force has been reached. Change from baseline in tactile response to Week 4 was calculated
Time Frame: Baseline to 4 weeks post administration of study treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | SnF Dentifrice | NaMFP Dentifrice
Number analyzed (Participants) | 60 | 58
grams | 11.2 (15.95) | 1.5 (3.86)
Statistical Analysis 1: Comparison: SnF Dentifrice vs NaMFP Dentifrice; Null hypothesis considered change from baseline to be same for both treatments; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment made for multiple comparisons, as primary comparison was pre-specified; ANCOVA with treatment as fixed factor and baseline Schiff Score as covariate; Adjusted Mean Difference = 9.6, 95% CI 2-sided [5.4 to 13.9] — Difference is 0.454% SnF minus 0.76% NaMFP such that a positive difference favors first named treatment

ADVERSE EVENTS:
Time Frame: All adverse events encountered or spontaneously reported following administration of any investigational product, or for up to 5 days after the last administration of investigational product were recorded.
Arm/Group | SnF Dentifrice | NaMFP Dentifrice
Serious Adverse Events (participants affected / at risk) | 0/60 | 1/58
Other Adverse Events (participants affected / at risk) | 1/60 | 0/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SnF Dentifrice (N=60) | NaMFP Dentifrice (N=58)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SnF Dentifrice (N=60) | NaMFP Dentifrice (N=58)
Oral Herpes (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.